CLINICAL TRIAL: NCT05471388
Title: Assessment of Serum Asprosin Level in Male Patients With Acne Vulgaris
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Esraa Abdel-Azeem Hamoda, resident doctor at Dematology, Venereology and Andrology department at Sohag University Hospital, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Soh-Med-22-07-06
Record Dates: First submitted 2022-07-20; First posted 2022-07-22 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Acne Vulgaris
Keywords: Asprosin
MeSH Terms: conditions — Acne Vulgaris; Arachnodactyly

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- case (Active Comparator)
  Interventions: Diagnostic Test: serum asprosin
- control (Active Comparator)
  Interventions: Diagnostic Test: serum asprosin

INTERVENTIONS:
Diagnostic Test: serum asprosin — assessment of serum asprosin by a commercially available double-antibody sandwich enzyme-linked immunosorbent assay (ELISA) kit.

SUMMARY:
Subject of interest is to evaluate serum level of asprosin in male patients with acne vulgaris, demonstrate the relation between acne vulgaris severity and level of asprosin in these patients & the relation between metabolic syndrome in acne vulgaris and level of asprosin.

ELIGIBILITY:
Inclusion Criteria:

* Acne vulgaris male patients (>18 years) will be included.

Exclusion Criteria:

* Age <18 years.
* Females.
* Patients with other inflammatory skin disorders.
* Patients with associated systemic diseases.
* Current or previous treatment with isotretinoin in the last 3 month ,anti-inflammatory drugs, systemic antibiotics, androgen or anti androgen therapy, and steroid therapy).
* Patients known on treatment of diabetes, hypertension and dyslipidemia.
* Athletes.
* Patient refusal.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — males
Enrollment: 72 (Estimated)
Dates: Start 2022-07-18 (Estimated); Primary Completion 2023-01-18 (Estimated); Study Completion 2023-01-18 (Estimated)

PRIMARY OUTCOMES:
Assess serum asprosin level in male patients with acne vulgaris. | 6 months
  Assess serum asprosin level in male patients with acne vulgaris.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Rocha MA, Bagatin E. Adult-onset acne: prevalence, impact, and management challenges. Clin Cosmet Investig Dermatol. 2018 Feb 1;11:59-69. doi: 10.2147/CCID.S137794. eCollection 2018. PMID 29440921
- [Background] Kovacs D, Fazekas F, Olah A, Torocsik D. Adipokines in the Skin and in Dermatological Diseases. Int J Mol Sci. 2020 Nov 28;21(23):9048. doi: 10.3390/ijms21239048. PMID 33260746
- [Background] Nagpal M, De D, Handa S, Pal A, Sachdeva N. Insulin Resistance and Metabolic Syndrome in Young Men With Acne. JAMA Dermatol. 2016 Apr;152(4):399-404. doi: 10.1001/jamadermatol.2015.4499. PMID 26720707
- [Background] Hong T, Li JY, Wang YD, Qi XY, Liao ZZ, Bhadel P, Ran L, Yang J, Yan B, Liu JH, Xiao XH. High Serum Asprosin Levels Are Associated with Presence of Metabolic Syndrome. Int J Endocrinol. 2021 Mar 2;2021:6622129. doi: 10.1155/2021/6622129. eCollection 2021. PMID 33747078